CLINICAL TRIAL: NCT07306052
Title: Safety and Efficacy of Epidural Spinal Cord Stimulation for Restoring Walking in Spinal Cord Injury
Brief Title: Epidural Spinal Cord Stimulation for Restoring Walking in Spinal Cord Injury
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Collaborators: Zhejiang University (Other)
Responsible Party: Principal Investigator, Junming Zhu, Chief Physician, Second Affiliated Hospital, School of Medicine, Zhejiang University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025-1940
Record Dates: First submitted 2025-12-12; First posted 2025-12-29 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Spinal Cord Injuries (SCI)
Keywords: Epidural Electrical Stimulation; Spincal cord stimulation; Spincal cord injury
MeSH Terms: conditions — Spinal Cord Injuries | interventions — Rehabilitation; Evoked Potentials, Somatosensory; Evoked Potentials, Motor; Diffusion Tensor Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Epidural spinal cord stimulation + Standard Rehabilitation (Experimental): Participants receive the epidural spnial cord stimulation combined with individualized standard rehabilitation therapy for 12 months.
  Interventions: Procedure: Epidural spinal cord stimulation; Procedure: Rehabilitation Therapy; Radiation: positron emission tomography-computed tomography (PET-CT); Procedure: Somatosensory Evoked Potentials (SEPs); Procedure: Motor Evoked Potentials (MEPs); Radiation: Diffusion Tensor Imaging (DTI)

INTERVENTIONS:
Procedure: Epidural spinal cord stimulation — Epidural spinal cord stimulation is a medical technology that involves delivering controlled electrical impulses to the spinal cord through electrodes implanted in the epidural space-the area between the outermost membrane of the spinal cord (dura mater) and the vertebrae. This technique aims to modulate the activity of spinal neural networks, thereby regulating neurological functions and promoting functional recovery, particularly in individuals with spinal cord injuries or certain neurological disorders.
Procedure: Rehabilitation Therapy — A structured, multidisciplinary rehabilitation program designed to improve motor function, mobility, and independence in participants with paralysis. The therapy typically includes physical Therapy and occupational Therapy.
Radiation: positron emission tomography-computed tomography (PET-CT) — PET-CT is an advanced hybrid imaging modality that combines metabolic information from positron emission tomography with anatomical details from computed tomography.
Procedure: Somatosensory Evoked Potentials (SEPs) — SEPs are electrophysiological responses recorded from the central or peripheral nervous system following electrical stimulation of sensory nerves. They assess the functional integrity of somatosensory pathways.
Procedure: Motor Evoked Potentials (MEPs) — MEPs are electrophysiological responses elicited by transcranial magnetic stimulation or electrical stimulation of the motor cortex, recorded from peripheral muscles or the spinal cord. They evaluate the integrity of corticospinal tracts.
Radiation: Diffusion Tensor Imaging (DTI) — DTI is an advanced MRI technique that maps white matter tracts by measuring the directionality (anisotropy) and magnitude of water molecule diffusion in neural tissues. It provides quantitative metrics of fibers.

SUMMARY:
The goal of this clinical trial is to evaluate the safety and effectiveness of Epidural Electrical Stimulation (EES) combined with rehabilitation training for the reconstruction of walking in patients with chronic spinal cord injury (SCI) classified as AIS C-D. The main questions it aims to answer are:

Does the intervention of EES combined with rehabilitation significantly improve walking capacity? Is the combined intervention a safe approach for this patient population? Researchers will compare participants' functional assessments before EES implantation and at 1, 3, 6, 9, and 12 months post-implantation to evaluate the longitudinal effects. The primary assessments include the Walking Index for Spinal Cord Injury II (WISCI II), the 10-Meter Walk Test (10mWT), and the 6-Minute Walk Test (6minWT). Secondary outcome measures encompass the International Standards for Neurological Classification of Spinal Cord Injury (ISNCSCI), the Spinal Cord Independence Measure (SCIM III), the Functional Independence Measure (FIM), the Modified Ashworth Scale (MAS), the Penn Spasm Frequency Scale, and pain Visual Analogue Scale (VAS) scores. Neurophysiological and imaging evaluations, including electromyography (EMG), motor evoked potentials (MEPs), somatosensory evoked potentials (SEPs), and positron emission tomography-computed tomography (PET-CT), will be conducted preoperatively and at 6 months postoperatively to explore the mechanisms of neuroplasticity.

Participants will:

Undergo surgical implantation of an EES device. Receive personalized EES parameter programming combined with rehabilitation training (≥2 hours daily) post-operatively.

Complete a series of standardized functional and clinical outcome assessments at scheduled follow-up intervals.

Undergo scheduled neurophysiological and metabolic imaging studies. Report any adverse events throughout the study duration.

ELIGIBILITY:
Inclusion Criteria:

* Age between 16 and 65 years.
* Diagnosed with traumatic spinal cord injury for ≥ 6 months and ≤ 36 months.
* American Spinal Injury Association Impairment Scale (AIS) grade C-D.
* Spinal cord injury level above T10;
* Walking Index for Spinal Cord Injury II (WISCI II) score < 13.
* Completion of a standard conventional rehabilitation program prior to enrollment.
* Preserved upper limb function sufficient for self-propelling a manual wheelchair.
* Sitting balance grade ≥ 1.
* Ability to elicit clear electromyographic responses in lower limb muscles (e.g., rectus femoris, biceps femoris, gastrocnemius, tibialis anterior) upon transcutaneous electrical spinal cord stimulation at the T12-L1 vertebral levels.
* Willingness to voluntarily participate, and commitment to compliance with all necessary postoperative rehabilitation, assessments, and follow-up visits.

Exclusion Criteria:

* History of myocardial infarction or stroke within the past 6 months.
* Diagnosis of psychiatric disorders with active suicidal ideation or risk.
* Current pregnancy or planned pregnancy during the study period.
* Bleeding tendency or coagulopathy (prothrombin time ≥18 seconds).
* History of alcohol or substance abuse or dependence.
* Intellectual disability, cognitive impairment, or personality disorders.
* Other chronic medical conditions that may interfere with rehabilitation (e.g., unhealed severe fractures, hepatic or renal failure, severe anemia, etc.).
* Implantation of cardiac pacemakers, cardioverters, or defibrillators.
* Any other condition deemed inappropriate for participation by the investigators.

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2025-12-12 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Adverse Events (AEs) | Entire study period from implantation to the 13-month postoperative follow-up.
  The incidence, severity, and relationship to the intervention of all AEs . All AEs will be defined, recorded, and graded according to the International Council for Harmonisation Good Clinical Practice guidelines. Serious adverse events will be reported specifically based on established criteria. This assessment will comprehensively cover all safety concerns related to the surgical procedure (epidural stimulator implantation), the electrical stimulation itself (across various parameter sets).
WISCI II (Walking Index for Spinal Cord Injury II) | baseline, and 2, 4, 7, 13 monthes after surgery.
  The WISCI II evaluates walking ability in spinal cord injury patients. It has 21 levels (0-20), with scores based on mobility aids and assistance needed. A score of 0 means no walking; 20 indicates independent walking without aids.
Spinal Cord Independence Measure III (SCIM III) | baseline, and 2, 4, 7, 13 months after surgery
  SCIM III is a disease-specific, validated assessment tool designed to evaluate the functional independence of individuals with spinal cord injury in performing essential activities of daily living, self-care, mobility, and respiration/management. It is tailored to reflect the unique challenges and priorities of the SCI population.
  The SCIM III consists of 19 items across three subscales:
  Self-care subscale (0-20 points): Includes feeding, grooming, bathing, and dressing.
  Respiration and sphincter management subscale (0-40 points): Covers respiration, bladder management, and bowel management.
  Mobility subscale (0-40 points): Assesses mobility in room and toilet, indoors and outdoors mobility, and stair management.
  The total score ranges from 0 to 100 points, with higher scores indicating greater functional independence.

SECONDARY OUTCOMES:
International Standards for Neurological Classification of Spinal Cord Injury (ISNCSCI) | baseline, and 2, 4, 7, 13 monthes after surgery
  ISNCSCI is the most authoritative and widely used standard for evaluating neurological function after spinal cord injury, comprising:
  Motor Scores:
  Range:
  Upper limbs (C5-T1): 0-25 per limb (total 0-50) Lower limbs (L2-S1): 0-25 per limb (total 0-50) Total motor score: 0-100 points Higher scores indicate better motor function
  Sensory Scores:
  Light touch:
  0-2 points per dermatome (C2-S4/5) Total: 0-112 points
  Pinprick:
  0-2 points per dermatome (C2-S4/5) Total: 0-112 points Interpretation: Higher scores indicate better sensory preservation Neurological Level of Injury: determined by the most caudal segment
  ASIA Impairment Scale (AIS) Grading:
  A = Complete (no motor/sensory function in S4-S5) B = Sensory incomplete C = Motor incomplete (<50% key muscles strength ≥3/5 grade) D = Motor incomplete (≥50% key muscles strength ≥3/5 grade) E = Normal
Functional Independence Measure (FIM) | baseline, and 2, 4, 7, 13 months after surgery
  The Functional Independence Measure (FIM) is a widely used assessment tool designed to evaluate a person's functional status and level of independence in daily living activities, particularly among individuals with disabilities.
  FIM items are scored based on the level of assistance required to complete a task, ranging from 1 to 7 points per item.
  The FIM consists of 18 items across two domains: Motor domain (13 items): Includes activities such as eating, grooming, bathing, dressing, toileting, transfers (bed/chair, toilet, tub/shower), walking, and stair climbing. Cognitive domain (5 items): Covers communication (comprehension and expression) and social cognition (memory, problem-solving, and social interaction).
  The total score ranges from 18 to 126 points:
  ≤ 35 points: Severe dependence 36-89 points: Moderate dependence 90-119 points: Mild dependence 120-126 points: Functional independence
The 10-Meter Walk Test (10m-WT) | baseline, and 2, 4, 7, 10, 13 monthes after surgery
  10mWT is a widely used, objective performance-based assessment tool designed to evaluate short-distance walking speed and functional mobility in individuals with neurological impairments, including spinal cord injury.
  The time taken to walk the middle 6 meters is recorded in seconds.
The 6-Minute Walk Test (6min-WT) | baseline, and 2, 4, 7, 10, 13 monthes after surgery
  The 6min-WT is a widely used, objective performance-based assessment tool designed to evaluate submaximal exercise capacity, functional endurance, and walking distance in individuals with chronic cardiopulmonary or neurological conditions, including spinal cord injury.
  The participant is instructed to walk back and forth as far as possible within the 6-minute time period, at a self-selected pace that can be sustained throughout the test.
Modified Ashworth Scale (MAS) | baseline, and 2, 4, 7, 13 monthes after surgery
  MAS is a clinical tool used to assess muscle spasticity by grading resistance during passive movement. It scores from 0 (no tone increase) to 4 (rigid joint), with intermediate grades: 1 (slight resistance), 1+ (mild resistance through ≤50% ROM), 2 (marked resistance), and 3 (considerable resistance). Higher MAS scores (max=4) indicate worse outcomes, reflecting more severe spasticity that impairs mobility.
Penn | baseline, and 2, 4, 7, 13 months after surgery
  The Penn Scale is a specific assessment tool for measuring muscle spasticity. Scores range from 0 (no spasticity) to 4 (severe, rigid spasticity), with higher scores indicating more intense muscle stiffness and involuntary contractions.
Visual Analog Scale (VAS) Pain Score | baseline, and 2, 4, 7, 13 monthes after surgery
  The VAS Pain Score is a self-reported measure of pain intensity. It consists of a 10-cm horizontal line, anchored by "no pain" (0) on one end and "worst pain imaginable" (10) on the other. Patients mark the line to represent their current pain level, and the score is determined by measuring the distance from "no pain." It provides a simple, quick method to quantify subjective pain experiences, monitor fluctuations, and guide pain management strategies.

OTHER OUTCOMES:
Surface Electromyography (EMG) | baseline, and 7 monthes after surgery
  EMG is a non-invasive electrophysiological assessment tool designed to quantify the electrical activity and activation patterns of lower-limb muscles during specific volitional or task-related motor attempts.
  EMG recordings are obtained using surface electrodes placed over key lower-lild muscles. The root mean square amplitude of the signal during defined task epochs is measured in microvolts. Changes in EMG amplitude and temporal coordination provide an objective measure of muscle recruitment efficacy, spinal motor pool excitability, and the recovery of coordinated motor output following neuromodulation and rehabilitation.
Motor Evoked Potentials (MEPs) | baseline, and 7 monthes after surgery
  MEPs are neurophysiological responses elicited by transcranial magnetic stimulation, designed to assess the integrity and conductivity of the corticospinal tract.
  MEP latency and peak-to-peak amplitude are recorded from target lower-limb muscles using surface EMG. Latency reflects conduction time along the central motor pathway, while amplitude correlates with the number of synchronously activated motor units and the excitability of spinal motoneurons. Changes in these parameters serve as quantitative biomarkers for the functional reorganization and strengthening of descending supraspinal control after intervention.
Somatosensory Evoked Potentials (SEPs) | baseline, and 7 monthes after surgery
  SEPs are neurophysiological responses elicited by electrical stimulation of peripheral nerves, designed to evaluate the integrity of the dorsal column-medial lemniscus sensory pathway.
  SEP latency and amplitude are recorded over the scalp following tibial nerve stimulation. Prolonged latency or reduced amplitude indicates impaired conduction within the ascending sensory tracts. Serial measurements provide an objective assessment of the recovery or reorganization of afferent sensory input to the cortex, complementing clinical sensory examinations.
Spinal ¹⁸F-FDG PET-CT | baseline, and 7 monthes after surgery
  Spinal ¹⁸F-FDG PET-CT is a molecular imaging modality designed to quantify regional glucose metabolism, serving as an indicator of neuronal and glial metabolic activity.
  The standardized uptake value ratio is calculated for defined spinal cord segments relative to a reference region. Changes in FDG uptake reflect alterations in synaptic activity, inflammation, or tissue repair processes. This measure provides a unique in vivo biomarker for assessing metabolis neuroplasticity and the longitudinal changes in spinal cord circuitry activity in response to epidural stimulation and rehabilitation.

CONTACTS AND LOCATIONS:
Overall Officials: Junming Zhu, Principal Investigator — Second Affiliated Hospital, School of Medicine, Zhejiang University
Locations (1):
- Second Affiliated Hospital, School of Medicine, Zhejiang University, Hangzhou, Zhejiang, China